CLINICAL TRIAL: NCT01062893
Title: Effect of Epidural Saline on Duration and Spread of Subsequent Spinal Analgesia/Anesthesia Using a CSE Technique
Brief Title: Combined Spinal/Epidural (CSE) Saline Duration/Spread
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of subjects and manpower issues
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00009631
Record Dates: First submitted 2010-02-01; First posted 2010-02-04 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Labor Pain
Keywords: labor pain treatment; duration analgesia; Analgesic duration with normal saline injection.; Analgesic duration without normal saline injection
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0 mls saline injected (Placebo Comparator): NO SALINE INJECTED
  Interventions: Other: Sterile normal saline 0 mls
- 15 mls saline (Active Comparator): 15ML SALINE ADMINISTERED EPIDURALLY
  Interventions: Other: 15 mls sterile normal saline

INTERVENTIONS:
Other: Sterile normal saline 0 mls — at time of epidural needle placement there will not be any saline injected into the epidural space prior to placement of the spinal needle to administer the CSE dose of standard analgesic medications. Instead a pause will be done as by the investigator to maintain blind for the assessor.
  Arms: 0 mls saline injected
Other: 15 mls sterile normal saline — After the epidural needle is placed, 15 mls of sterile normal saline will be injected into the epidural space, then the spinal needle will be placed to administer the CSE dose of standard analgesic medications.
  Arms: 15 mls saline

SUMMARY:
An attempt is being made to see if by injecting a set volume of sterile saline into the epidural space during the treatment of labor pain with a combined spinal/epidural (CSE) increases the amount of pain relief obtained and makes the labor analgesia lasts longer. Subjects are in the study from the time their CSE is placed until they request additional pain medication from the spinal dose of numbing medicine wearing off.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 12 years of age
* ASA status 1 or 2
* cervical dilation < 6cm

Exclusion Criteria:

* ASA assigned 3 or 4
* advanced labor (> 6cm cervical dilated)
* distorted epidural anatomy

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Pan, MD, MSEE, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Forsyth Medical Center-Sara Lee Center for Women's Health, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Started | 41 | 41
Completed | 27 | 28
Not Completed | 14 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 28 | 55
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Highest Sensory Blockade Level to Pinprick and to Cold
Description: Onset of analgesia to recession of analgesia. Highest spread of analgesia (highest sensory level) to cold temp and pinprick, with level defined from T1 to L5, where T1 is highest =level 17 and L5 is lowest =Level 1)
Time Frame: up to 20 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 27 | 28
units on a scale | 10.1 (2.9) | 11.6 (1.9)

2. Secondary Outcome: Duration of Analgesia (Time to Request Additional Analgesia)
Description: time of CSE to time request of additional supplement analgesia in minutes
Time Frame: up 120 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 27 | 28
minutes | 57.2 (33.9) | 77.3 (30.0)

3. Secondary Outcome: Onset of Analgesia
Description: time to VAS</=3 on a 0-10 scale with 0=no pain up to 10= worst pain imaginable
Time Frame: up to 20 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 27 | 28
minutes | 7.96 (5.24) | 6.07 (3.15)

4. Secondary Outcome: Time to Highest Sensory Block
Time Frame: up to 20 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 27 | 28
minutes | 12.96 (8.69) | 13.57 (6.5)

5. Secondary Outcome: Number of Participants Who Had Occurrence of Fetal Bradycardia
Description: occurrence of common side effects of spinal/epidural administration
Time Frame: length of labor, up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 27 | 28
Participants | 1 | 0

6. Secondary Outcome: Number of Participants Who Had Occurrence of Maternal Hypotension
Time Frame: length of labor, up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 27 | 28
Participants | 2 | 4

7. Secondary Outcome: Occurrence of Use of Vasopressors
Time Frame: length of labor, up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 27 | 28
Participants | 10 | 12

8. Secondary Outcome: Number of Participants Who Had Occurrence of Itching
Time Frame: length of labor, up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 27 | 28
Participants | 1 | 1

9. Secondary Outcome: Number of Participants Who Had Occurrence of Post Dural Puncture Headache
Time Frame: length of labor, up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 27 | 28
Participants | 0 | 0

10. Secondary Outcome: Time for 2 Dermatome Level Regression of Sensory Block
Time Frame: up to 20 minutes
Population: No data collected
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time for Regression of Motor Blockade
Time Frame: up to 20 minutes
Population: No data collected
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | 0 Mls Saline Injected | 15 Mls Saline
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-01-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT01062893/Prot_SAP_000.pdf